CLINICAL TRIAL: NCT00680693
Title: Mindfulness for Irritable Bowel Syndrome
Brief Title: Mindfulness vs. Support Groups for Irritable Bowel Syndrome
Acronym: M-IBS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Susan Gaylord, Assistant Professor, University of North Carolina, Chapel Hill
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R21AT003619-02 (NIH); R21AT003619-02 (NIH)
Record Dates: First submitted 2008-05-15; First posted 2008-05-20 (Estimated); Last update posted 2011-11-18 (Estimated); Status verified 2010-02

CONDITIONS: Irritable Bowel Syndrome
Keywords: IBS, functional gastrointestinal disease
MeSH Terms: conditions — Irritable Bowel Syndrome; Ichthyosis Bullosa of Siemens

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Mindfulness-based stress management 8-week program
  Interventions: Behavioral: Mindfulness training
- 2 (Active Comparator): Psycho-educational support group for women with IBS
  Interventions: Behavioral: Psycho-educational support group for women with IBS

INTERVENTIONS:
Behavioral: Mindfulness training — 8 weekly 2-hour classes
  Arms: 1
Behavioral: Psycho-educational support group for women with IBS — 8 weekly 2-hour meetings
  Arms: 2

SUMMARY:
Irritable bowel syndrome (IBS) is a common and disabling functional disorder characterized by significant abdominal discomfort and disturbed defecation. It affects over 10% of U.S. adults (14% women, 8% men), resulting in major disability, impaired quality of life, and a significant health-care burden. Conventional management of IBS is only partially effective in some patients and includes use of medications, behavioral modification, dietary approaches, and lifestyle changes such as exercise and stress reduction. Although behavioral treatments such as cognitive behavioral therapy and hypnosis have been among the most effective treatments, they are costly to deliver.

Mindfulness meditation, a complementary/alternative medicine (CAM) therapy taught in groups, is a unique self-regulatory, mind-body approach in which practitioners learn to attend to present-moment experiences, letting go of fixation on negative emotions and thoughts of past and future. It has been found to be effective in reducing chronic pain and stress and in ameliorating disorders with similarities to IBS, including fibromyalgia, headache, and depression.

The overall goals of this exploratory, pilot study of women with IBS are to compare mindfulness meditation training to a patient support group (a previously validated control condition) in a small, randomized controlled clinical trial, in order to assess the feasibility of a larger, definitive trial. Specific aims are to evaluate primary and secondary outcome measures, to assess expectancy of benefit and scales measuring mindfulness (process measures), and to identify barriers to conducting such a trial in our setting. Sixty women meeting Rome II diagnostic criteria for IBS will be randomly assigned to one of two treatments - mindfulness meditation training or a support group - and will undergo 8 weekly group sessions plus a single day-long session. The primary outcome measure is improvement on the validated Irritable Bowel Symptom Severity Scale from pretreatment to the end of treatment, with follow-up at 3, 6, and 12 months. Additional variables address alternative endpoints (e.g., Adequate Relief of IBS symptoms, disease specific quality of life) and mechanism of treatment effects (e.g., coping scales, psychological symptoms, Visceral Sensitivity Scale). The multidisciplinary research team includes physicians, psychologists, and educators.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older, female, English-speaking, confirmed IBS meeting Rome II criteria with a minimum duration of symptoms of six months and under the care of a physician for IBS; able to provide informed consent; willing and able to document IBS symptoms and use of medications, as well as complete the assessment instruments. Subjects must be willing to attend and participate in 8 weekly Mindfulness Program or Support Group sessions.

Exclusion Criteria:

* Evidence of severe neuropsychological impairment or psychosis, significant depression, anxiety, a history of an inpatient admission for psychiatric disorder within the past two years; pregnancy or anticipated pregnancy; undergoing active treatment for a major medical illness such as malignancy, diabetes, autoimmune or immune deficiency disorder; a history of inflammatory bowel disease, gastrointestinal malignancy, active liver or pancreatic disease including diabetes, uncontrolled lactose intolerance, celiac disease, a history of abdominal trauma or surgery, cognitive impairment that prevents understanding or responding to study questions; prior history of mindfulness meditation training. Given the highly verbal nature of the interventions, otherwise eligible patients who do not speak or write English will be excluded from this study.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Actual)
Dates: Start 2006-10; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

PRIMARY OUTCOMES:
IBS-S | 3 months

SECONDARY OUTCOMES:
Visceral Sensitivity Index | 3 months
Work Productivity and Activity Impairment for IBS (WPAI:IBS) | 3 months
Recent Physical Symptoms Questionnaire (RPSQ) | 3 months
Brief Symptom Inventory (BSI) | 3 months
State Trait-Anger Expression Inventory (STAXI) | 3 months
Coping Strategies Questionnaire (CSQ) | 3 months
IBS QOL | 3 months
Daily Symptom Diary | Daily x 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Susan A Gaylord, PhD, Principal Investigator — University of North Carolina, Chapel Hill
Locations (1):
- University of North Carolina at Chapel Hill, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Gaylord SA, Whitehead WE, Coble RS, Faurot KR, Palsson OS, Garland EL, Frey W, Mann JD. Mindfulness for irritable bowel syndrome: protocol development for a controlled clinical trial. BMC Complement Altern Med. 2009 Jul 28;9:24. doi: 10.1186/1472-6882-9-24. PMID 19638214